CLINICAL TRIAL: NCT02312245
Title: Avatar-Directed Chemotherapy in Platinum-Resistant Ovarian, Primary Peritoneal and Fallopian Tube Cancers
Brief Title: Avatar-Directed Chemotherapy in Treating Patients With Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1463; NCI-2014-02399 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14-002986 (Other: Mayo Clinic Institutional Review Board); MC1463 (Other: Mayo Clinic); R01CA184502 (NIH)
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Gemcitabine; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (Avatar-directed paclitaxel) (Experimental): Patients receive paclitaxel IV over 1-96 hours on days 1, 8, and 15. Patients may also receive bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: Bevacizumab; Drug: Paclitaxel
- Arm B (Avatar-directed gemcitabine hydrochloride) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride
- Arm C (Avatar-directed liposomal doxorubicin) (Experimental): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1. Patients may also receive bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Pegylated Liposomal Doxorubicin Hydrochloride
- Arm D (Avatar-directed topotecan hydrochloride) (Experimental): Patients receive topotecan hydrochloride IV over 30 minutes on days 1-5 every 21 days or days 1, 8, and 15 every 28 days. Patients may also receive bevacizumab IV over 90 minutes on day 1 every 21 days or days 1 and 15 every 28 days. Courses repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm A (Avatar-directed paclitaxel); Arm C (Avatar-directed liposomal doxorubicin); Arm D (Avatar-directed topotecan hydrochloride)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
  Arms: Arm B (Avatar-directed gemcitabine hydrochloride)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm A (Avatar-directed paclitaxel)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; DOX-SL; Doxil; Doxilen; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm C (Avatar-directed liposomal doxorubicin)
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm D (Avatar-directed topotecan hydrochloride)

SUMMARY:
This phase II trial studies how well Avatar-directed chemotherapy works in treating patients with ovarian, primary peritoneal, or fallopian tube cancer that does not respond to platinum anti-cancer drugs. Drugs used in chemotherapy, such as paclitaxel, gemcitabine hydrochloride, pegylated liposomal doxorubicin hydrochloride, topotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Using an Avatar, a living tumor sample with similar genetic characteristics to the original tumor, may help determine which chemotherapy is most effective.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate of Avatar-directed salvage chemotherapy in patients with platinum-resistant ovarian, primary peritoneal and fallopian tube cancers.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival of patients with platinum-resistant ovarian, primary peritoneal and fallopian tube cancers receiving Avatar-directed salvage chemotherapy.

II. To determine the overall survival of patients with platinum-resistant ovarian, primary peritoneal and fallopian tube cancers receiving Avatar-directed salvage chemotherapy.

III. To determine the adverse events for patients with platinum-resistant ovarian, primary peritoneal and fallopian tube cancers receiving Avatar-directed salvage chemotherapy.

IV. To determine the correlation between patient response and response in their Avatar.

V. To enrich the Avatar response signature in response to Avatar-directed therapy using patient outcomes.

VI. To compare the response rates between patients who did or did not receive bevacizumab treatment.

OUTLINE: Patients are assigned to 1 of 4 treatment arms as directed by Avatar results.

ARM A: Patients receive paclitaxel intravenously (IV) over 1-96 hours on days 1, 8, and 15. Patients may also receive bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity

ARM B: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1. Patients may also receive bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive topotecan hydrochloride IV over 30 minutes on days 1-5 every 21 days or days 1, 8, and 15 every 28 days. Patients may also receive bevacizumab IV over 90 minutes on day 1 every 21 days or days 1 and 15 every 28 days. Courses repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of ovarian, primary peritoneal or fallopian tube cancer of any subtype
* Prior consent to have tumors used for unspecified future research
* Ability to provide written informed consent
* Willing to agree to periodic contact with a member of the study team during the period that the cancer has not recurred and/or has not become platinum resistant
* Willing to agree that the local medical oncologist may be informed that patient has agreed to participate in the study
* Platinum resistant or refractory ovarian, primary peritoneal or fallopian tube cancer of any subtype; Note: platinum-sensitive disease is allowed in cases where there is a contraindication to platinum-based therapy (i.e., allergy to platinum); this must be reviewed and approved by the Principal Investigator
* Successful Avatar engraftment with successful expansion and treatment outcome of Avatar therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (ECOG performance status [PS]) of 0, 1 or 2
* Measurable disease or non-measurable disease; for patients with non-measureable disease, they must also have a cancer antigen (CA)-125 measurement of > 35 U/mL or 2 X their documented nadir on 2 separate measurements 1 week apart
* The following laboratory values obtained =< 21 days prior to registration; complete blood count (CBC), sodium, potassium, aspartate aminotransferase (AST), bilirubin and creatinine are to be obtained pre-study; Note: treatment initiation and dosing modification should be performed at the individual investigators discretion and be consistent with the product label and their medical practice
* Negative urine or serum pregnancy test performed =< 7 days prior to registration, for women of child bearing potential only
* Willing to return to enrolling institution for follow-up or have a local physician willing to submit response and outcome data; Note: any and all therapy, potentially in its entirety, may be conducted outside of the Mayo Clinic

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
* Prior treatment with Doxil, topotecan, Gemzar or Taxol chemotherapy for platinum-resistant cancer; Note: Allowed prior therapy with Doxil or Gemzar if given for platinum sensitive disease in combination with a platinum drug AND the Avatar data indicates a drug other than Doxil or Gemzar would be effective; Note: Allowed prior therapies for patients following confirmation of platinum-resistant cancer include:

  * Therapeutic antibodies, such as bevacizumab
  * Small molecule kinase inhibitors, such as pazopanib
  * Vaccines and immunotherapy All of these exceptions should be confirmed with the Principal Investigator (PI) prior to registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; Note: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness judged by the treating investigator to preclude treatment with chemotherapy
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; Note: if there is a history of prior malignancy, they must not be receiving treatment for their cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Weroha, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Avatar-directed Paclitaxel): Patients receive paclitaxel IV over 1-96 hours on days 1, 8, and 15. Patients may also receive bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity> > Bevacizumab: Given IV>
  > Paclitaxel: Given IV
- Arm B (Avatar-directed Gemcitabine Hydrochloride): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  > Gemcitabine Hydrochloride: Given IV
- Arm C (Avatar-directed Liposomal Doxorubicin): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 60 minutes on day 1. Patients may also receive bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.> > Bevacizumab: Given IV>
  > Pegylated Liposomal Doxorubicin Hydrochloride: Given IV
- Arm D (Avatar-directed Topotecan Hydrochloride): Patients receive topotecan hydrochloride IV over 30 minutes on days 1-5 every 21 days or days 1, 8, and 15 every 28 days. Patients may also receive bevacizumab IV over 90 minutes on day 1 every 21 days or days 1 and 15 every 28 days. Courses repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.> > Bevacizumab: Given IV>
  > Topotecan Hydrochloride: Given IV
Period: Overall Study
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm C (Avatar-directed Liposomal Doxorubicin) | Arm D (Avatar-directed Topotecan Hydrochloride)
Started | 3 | 1 | 0 | 9
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 0 | 9
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2
Not completed — Alternative Therapy | 1 | 0 | 0 | 0
Not completed — Progression | 0 | 0 | 0 | 5
Not completed — Patient went to hospice | 0 | 0 | 0 | 1
Not completed — Ineligible | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were enrolled were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm C (Avatar-directed Liposomal Doxorubicin) | Arm D (Avatar-directed Topotecan Hydrochloride) | Total
Number analyzed (Participants) | 3 | 1 | 0 | 9 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.54) | 32 (NA) — SD cannot be calculated for 1 patient |  | 56.6 (8.22) | 55.7 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 |  | 9 | 13
  Male | 0 | 0 |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0 | 0
  Not Hispanic or Latino | 3 | 1 |  | 9 | 13
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0
  Asian | 0 | 0 |  | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0
  Black or African American | 0 | 0 |  | 0 | 0
  White | 3 | 1 |  | 8 | 12
  More than one race | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 |  | 9 | 13
Tumor Histology Type [Count of Participants; unit: Participants]
  Ovarian (serous) | 3 | 1 |  | 7 | 11
  Fallopian tube (serous) | 0 | 0 |  | 1 | 1
  Ovarian (other) | 0 | 0 |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Confirmed Tumor Response, Defined as Complete Response or Partial Response Estimated Using Response Evaluation Criteria in Solid Tumors 1.1 Criteria
Description: Estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the exact Binomial method. The primary analysis will pool across all patients, and tumor response rate by treatment arm will also be looked at in an exploratory fashion.
Time Frame: 24 weeks
Population: All patients that were eligible and began treatment were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Avatar-directed Paclitaxel): Patients receive paclitaxel IV over 1-96 hours on days 1, 8, and 15. Patients may also receive bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity >
  > Bevacizumab: Given IV
  >
  > Paclitaxel: Given IV
- Arm B (Avatar-directed Gemcitabine Hydrochloride): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Gemcitabine Hydrochloride: Given IV
- Arm D (Avatar-directed Topotecan Hydrochloride): Patients receive topotecan hydrochloride IV over 30 minutes on days 1-5 every 21 days or days 1, 8, and 15 every 28 days. Patients may also receive bevacizumab IV over 90 minutes on day 1 every 21 days or days 1 and 15 every 28 days. Courses repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Bevacizumab: Given IV
  >
  > Topotecan Hydrochloride: Given IV
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm D (Avatar-directed Topotecan Hydrochloride)
Number analyzed (Participants) | 2 | 1 | 9
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Patients Experiencing Grade 3+ Adverse Events (AE)
Description: Maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine AE patterns.
Time Frame: 9 months
Population: All patients that were eligible and began treatment were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm D (Avatar-directed Topotecan Hydrochloride)
Number analyzed (Participants) | 2 | 1 | 9
Participants | 1 | 1 | 4

3. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated using the method of Kaplan-Meier. Analysis will be conducted with all arms of Avatar-directed chemotherapy pooled.
Time Frame: 25 months
Population: All patients that were eligible and began treatment were analyzed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm D (Avatar-directed Topotecan Hydrochloride)
Number analyzed (Participants) | 2 | 1 | 9
months | 7.9 [NA to NA] — The confidence interval was not able to be estimated due to a low number of events | 8.7 [NA to NA] — The confidence interval was not able to be estimated due to a low number of events | 9.2 [4.5 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS will be estimated using the method of Kaplan-Meier. Analysis will be conducted with all arms of Avatar-directed chemotherapy pooled.
Time Frame: 9 months
Population: All patients that were eligible and began treatment were analyzed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm D (Avatar-directed Topotecan Hydrochloride)
Number analyzed (Participants) | 2 | 1 | 9
months | 7.9 [NA to NA] — The confidence interval was not able to be estimated due to a low number of events | 8.7 [NA to NA] — The confidence interval was not able to be estimated due to a low number of events | 3.0 [1.9 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events

5. Secondary Outcome: Number of Patients With a Partial or Confirmed Response
Description: The Chi-square or Fisher's Exact test will be used to compare the response rates between patients who did or did not receive bevacizumab treatment. The response rates will also be reported by treatment type.
Time Frame: 9 months
Population: All patients that were eligible and began treatment were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm D (Avatar-directed Topotecan Hydrochloride)
Number analyzed (Participants) | 2 | 1 | 9
Participants | 0 | 0 | 0

6. Other Pre Specified Outcome: Enriched Avatar Response Signature in Response to Avatar-directed Therapy Using Patient Outcomes
Description: This will be an exploratory analysis that will use the outcome data from this trial to inform future work using Avatar directed therapy.
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Frequency (%) of Patients Who Had an Avatar Response and a Clinical Tumor Response for the Same Treatment
Description: Overall concordance rate and confidence interval will be reported.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 25 months
Arm/Group | Arm A (Avatar-directed Paclitaxel) | Arm B (Avatar-directed Gemcitabine Hydrochloride) | Arm D (Avatar-directed Topotecan Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/1 | 6/9
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 3/9
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Avatar-directed Paclitaxel) (N=2) | Arm B (Avatar-directed Gemcitabine Hydrochloride) (N=1) | Arm D (Avatar-directed Topotecan Hydrochloride) (N=9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Avatar-directed Paclitaxel) (N=2) | Arm B (Avatar-directed Gemcitabine Hydrochloride) (N=1) | Arm D (Avatar-directed Topotecan Hydrochloride) (N=9)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT02312245/Prot_SAP_000.pdf